CLINICAL TRIAL: NCT05402046
Title: A Multicentre, Prospective, Low-intervention Clinical Trial to Validate a Mobile Application ("ProRodinki") in Assessing the Risk of Skin Malignancies
Brief Title: Clinical vAlidation of a MobilE appLication ("ProRodinki") in the Assessment of the maLignant skIn neoplAsms
Acronym: CAMELLIA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: MelanomaPRO, Russia (Other)
Collaborators: Privolzhsky Research Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MELPRO-0821
Record Dates: First submitted 2022-05-29; First posted 2022-06-02 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: Melanoma (Skin); Nevus; Nevus, Spitz; Nevus Halo; Nevus, Pigmented; Basal Cell Carcinoma; Squamous Cell Carcinoma; Bowen's Disease; Melanoma in Situ; Spot Pigmented
MeSH Terms: conditions — Melanoma; Nevus; Nevus, Epithelioid and Spindle Cell; Nevus, Halo; Nevus, Pigmented; Carcinoma, Basal Cell; Carcinoma, Squamous Cell; Bowen's Disease

STUDY DESIGN:
Intervention Model Description: This is a multicentre, low-intervention, prospective study. Patients scheduled for excisional biopsy of skin lesion(s) will be invited to participate in this study. Photo-documentation of the skin neoplasm(s) in the ProRodinki application will be performed, and the generated report will be sent for evaluation by artificial intelligence. Following this procedure, an excisional biopsy of the lesion(s) will be scheduled. From the moment of inclusion in the study until the excisional biopsy, an interval of no more than 2-4 weeks is allowed. After excisional biopsy of the skin neoplasm(s), a routine intravital pathological examination with hematoxylin and eosin staining will be performed, if necessary, immunohistochemical and molecular genetic tests will be performed. The selected biosamples (paraffin blocks) will then be analyzed centrally by a morphologist.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ProRodinki application test (Experimental): Patients scheduled for excisional biopsy of skin lesion(s) will be invited to participate in this study. Photo-documentation of the skin neoplasm(s) in the ProRodinki application will be performed, and the generated report will be sent for evaluation by artificial intelligence. Following this procedure, an excisional biopsy of the lesion(s) will be scheduled. From the moment of inclusion in the study until the excisional biopsy, an interval of no more than 2-4 weeks is allowed. After excisional biopsy of the skin neoplasm(s), a routine intravital pathological examination with hematoxylin and eosin staining will be performed, if necessary, immunohistochemical and molecular genetic tests will be performed. The selected biosamples (paraffin blocks) will then be analyzed centrally by a morphologist.
  Interventions: Other: Mobile phone application "ProRodinki"

INTERVENTIONS:
Other: Mobile phone application "ProRodinki" — Patient were underwent photography using mobile phone and tested application "ProRodinki"just before preplanned excisional or incisional biopsy.
  Application AI result than will be compared with pathology report by independent investigator

SUMMARY:
A Multicenter, Prospective, Low-interventional Clinical Study Evaluating on mobile application validation ("ProRodinki") in assessing the risk of skin malignant neoplasms

DETAILED DESCRIPTION:
This is a multicentre, low-intervention, prospective study. In several centers, patients will be selected into 4 cohorts:

1. Patients with complaints of skin neoplasm(s) who have sought the help of a specialist to remove it(them), and patients with an established clinical diagnosis of suspicious/doubtful skin neoplasm(s) who are scheduled to undergo excisional biopsy to verify the diagnosis;
2. Patients who have complaints about a skin neoplasm(s) and consider it (them) suspicious without using the ProRodinki application and who have asked for help from a specialist in order to remove it(them);
3. patients who have complaints about skin neoplasm(s) and who, using the ProRodinki application, received a response that the neoplasm(s) is (are) suspicious / doubtful (s), and sought help from a specialist in order to remove it (their) to verify the diagnosis;
4. Cohort 4 (prospective): patients with suspicious/doubtful skin neoplasm(s) detected during an objective examination by a specialist without using the ProRodinki application, and who are scheduled for an excisional biopsy to verify the diagnosis .

Patients scheduled for excisional biopsy of skin lesion(s) will be invited to participate in this study. After signing the informed voluntary consent form in the ProRodinki application, an account will be created for the patient, in which a questionnaire will be filled out, photo-documentation of the skin neoplasm(s) will be performed, and the generated report will be sent for evaluation by artificial intelligence. The response received from the application for each clinical case will be recorded and all neoplasms will be grouped according to the classification of the application. Following this procedure, an excisional biopsy of the lesion(s) will be scheduled. From the moment of inclusion in the study until the excisional biopsy, an interval of no more than 2-4 weeks is allowed. Immediately before the excisional biopsy procedure, other non-invasive instrumental examinations (dermatoscopy, digital dermatoscopy) will be performed. After excisional biopsy of the skin neoplasm(s), a routine intravital pathological examination with hematoxylin and eosin staining will be performed, if necessary, immunohistochemical and molecular genetic tests will be performed. The selected biosamples (paraffin blocks) will then be analyzed centrally by a morphologist. All neoplasms will be classified according to the MPATH-Dx classification, the 2018 WHO classification of skin tumors, and will be assigned an ICD-O-3 code. For invasive melanomas, the characteristics necessary to establish the morphological stage of pT will also be collected (see also the Study Procedures section). The conclusion of the intravital pathoanatomical examination will be photo-documented through the ProRodinki application and attached to the patient's account in the tab where the photo of the removed neoplasm is stored.

ELIGIBILITY:
Inclusion Criteria:

General (for all cohorts):

* Signed informed consent form for participation in the study;
* Age of the patient over 18 years of age at the time of inclusion in the study (at the time of signing the consent form).
* The patient is scheduled for an incisional/excisional biopsy (or wide excision) of the skin lesion(s) within 2-4 weeks from entry into the study and the patient is able to tolerate this intervention;

Cohort 1 (prospective): Patients complaining of a skin lesion(s) who sought specialist help to remove it(s) and patients with a clinical diagnosis of suspicious/doubtful skin lesion(s) who are scheduled for excisional biopsy to verify the diagnosis

1. Patients who have complaints about skin neoplasm(s) and who have sought the physician to remove it(them);
2. Clinically suspicious/doubtful skin neoplasm(s) detected during an objective examination by a dermatologist or oncologist without the use of instrumental diagnostic methods;

Cohort 2 (prospective): Patients who complain of a skin neoplasm(s) and consider it(them) suspicious without using the ProRodinki application and seek specialist help to remove it(them)

1. Patients who have complaints about a skin neoplasm(s) and consider it (them) suspicious without using the ProRodinki application and who have asked a physician to remove it(them);
2. Clinically suspicious/doubtful skin neoplasm(s) detected during an objective examination by the patient without using the ProRodinki application;

Cohort 3 (prospective): patients who complained of skin neoplasm(s) and who, using the ProRodinki application, received an answer that the neoplasm(s) is (are) suspicious/doubtful(s), and applied for help from a specialist in order to remove it (their) to verify the diagnosis

1. Patients who have complaints about skin neoplasm(s), and who, using the ProRodinki application, received a response that the neoplasm(s) is (are) suspicious / doubtful (s), and referred to the physician to remove it (their) to verify the diagnosis;
2. Clinically suspicious/doubtful skin neoplasm(s) detected by the patient when using the ProRodinki application;

Cohort 4 (prospective): patients with suspicious/doubtful skin neoplasm(s) detected during an objective examination by a specialist without using the ProRodinki app, and who are scheduled for an excisional biopsy to verify the diagnosis

1. Patients who have a suspicious/dubious skin neoplasm(s) detected during an objective examination by a specialist without using the ProRodinki application, and who are scheduled to undergo an excisional biopsy to verify the diagnosis;
2. Clinically suspicious(s)/doubtful(s) skin neoplasm(s) detected during an objective examination by a dermatologist or oncologist without the use of instrumental diagnostic methods and the ProRodinki application;

Exclusion Criteria:

General (all cohorts):

* Patient is NOT scheduled for excisional biopsy (or wide excision) of skin lesion(s) within 3 months of enrollment in the study OR the patient is unable to tolerate this intervention;
* Available intravital pathological confirmation of the nature of the neoplasm(s) (benign or malignant) that(s) are planned to be removed as part of this study;
* Neoplasm(s) located subcutaneously or in soft tissues and, according to clinical signs, having no connection with the skin;
* Allergic reaction to drugs used during incisional / excisional biopsy or wide excision;
* The patient's inability to follow study procedures (including contact with the investigator during observation visits) or other reasons that, in the opinion of the principal investigator, may become an obstacle to the patient's participation in the study;
* For the period of inclusion in the study, do not sign the informed consent form;
* The age of the patient is younger than 18 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 605 (Estimated)
Dates: Start 2022-04-23 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Sensitivity for malignant neoplasm 90% or higher | 12 months
  Sensitivity will be calculated as the number of malignant neoplasms that are correctly classified, divided by all excised malignant neoplasms according to pathology report

CONTACTS AND LOCATIONS:
Overall Officials: Lev V Demidov, Professor, Study Director — The Russian Melanoma Professional Association (Melanoma.PRO); Igor V Samoylenko, Study Chair — The Russian Melanoma Professional Association (Melanoma.PRO)
Locations (2):
- Russia (2):
  - N.N.Blokhin Russian Cancer Research Center, Moscow
  - Privolzhsky Research Medical Unversity, Nizhny Novgorod

IPD SHARING:
Plan to Share IPD: Undecided